CLINICAL TRIAL: NCT05550584
Title: High Flow Oxygen During ProcEdural Sedation for Operative Hysteroscopy: a Randomized Controlled Trial - HOPE Study.
Brief Title: High Flow Oxygen During Operative Hysteroscopy.
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4872
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2022-07

CONDITIONS: Endometrium; Hypertrophy, Cervix; Anesthesia; Apnea, Postanesthetic
Keywords: High flow nasal cannula Oxygen; Procedural sedation; Apnoeic ventilation; Operative hysteroscopy; THRIVE
MeSH Terms: conditions — Hypertrophy; Butyrylcholinesterase deficiency | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (Experimental): Ventilatory management during surgery provided by transnasal humidified rapid-insufflation ventilatory exchange.
  Interventions: Device: Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE).
- Control (Active Comparator): Ventilatory management during surgery provided by mechanical ventilation through laringeal mask
  Interventions: Device: LMA

INTERVENTIONS:
Device: Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE). — In the THRIVE group, dedicated Optiflow THRIVE nasal cannulas will be positioned for 100% high flow oxygen therapy at an initial flow of 30 L/min. After induction of anesthesia and throughout the procedure the flow of oxygen will be increased to 70 L/min.
  Arms: THRIVE
Device: LMA — Mechanical ventilation performed by a laringeal mask
  Arms: Control

SUMMARY:
High-flow nasal cannula (HFNC) oxygen therapy represents an open circuit ventilation system that uses flows up to 70 L/min of 100% oxygen through the Optiflow THRIVETM device (Fisher and Paykel Healthcare Ltd, Auckland, New Zealand). Compared to conventional oxygen therapy systems, the heating and humidification of the flows facilitate tolerability by the patient, allow to reach higher and more stable inspiratory fractions of oxygen, produce a flow-dependent effect of continuous positive airway pressure and by reducing dead space, have the potential to increase alveolar volume and improve gas exchanges.

The use of HFNC is increased in anesthesia as the only airways management technique during short-term procedures under procedural sedation or general anesthesia.

Operative hysteroscopy is a short-term procedure (<30 minutes), usually performed in a day-hospital regimen, under procedural sedation. In case of apnea and/or hypoventilation, or for long and complex hysteroscopic procedures, the patient can be ventilated through facial or laryngeal masks.

The primary objective of this prospective randomized controlled trial is to compare the rate of success of ventilation using the THRIVE device to laryngeal mask ventilation during operative hysteroscopies under procedural sedation.

Secondary objectives will be the comparison of the percentage of complications in terms of inability to manage the airways, episodes of hypotension, cardiac arrhythmias, post-operative nausea and vomiting, degree of dyspnea and comfort of the patient in the Post-Anesthesia Care Unit between the two methods.

DETAILED DESCRIPTION:
High-flow nasal cannula (HFNC) oxygen therapy represents an open circuit ventilation system that uses flows up to 70 L/min of 100% oxygen through Optiflow THRIVETM (transnasal humidified rapid-insufflation ventilatory exchange) device (Fisher and Paykel Healthcare Ltd, Auckland, New Zealand).

Compared to conventional low-flows oxygen therapy systems, the heating and humidification of the flow facilitate tolerability by the patient, ensure an efficient muco-ciliary function and allow to reach higher and more stable inspiratory fractions of oxygen.

The system produces a flow-dependent effect of continuous positive airway pressure of about 1 cmH20 for every 10L/min increase in oxygen flow and a reduction of the dead space, having the potential to increase the alveolar volume thus improving gas exchanges.

The resulting reduction in respiratory rate and the improvement of thoracoabdominal synchrony minimize the onset of respiratory fatigue in the patient.

Initially introduced for the treatment of acute hypoxemic respiratory failure, HFNC oxygen therapy is increasingly used also in anesthesia as the only airways management technique during short-term procedures performed under sedation (e.g. digestive endoscopy) or under general anesthesia (such as microlaryngoscopies).

Compared to low-flows oxygen systems, the greater CO2 elimination capacity could reduce the incidence of hypoventilation and apnea episodes potentially associated with patient sedation.

Operative hysteroscopy is a brief procedure, normally lasting <30 minutes, usually performed in a day-hospital regime under procedural analgo-sedation, with conventional ventilatory support through a face mask/laryngeal mask.

The primary objective of this study is the comparison of the rate of success in airways management via the THRIVE system versus positive pressure ventilation by I-gel laryngeal mask during 180 hysteroscopies performed under general anesthesia.

Secondary objectives are: the comparison of intraoperative and postoperative complications between the two groups.

Materials and methods Patient monitoring throughout the procedure will include automatic noninvasive, intermittent (every 5 minutes) blood pressure monitoring, 3-leads electrocardiogram, peripheral oxygen saturation (SpO2), bispettral index (BIS), transcutaneous capnography with TCM5 Radiometer monitor.

Upon arrival in the operating room, the patient will assume the lithotomic position; a peripheral venous cannula will be placed at the level of the hand or forearm and it will begin the infusion of Ringer Lactate solution 3 ml/kg/h. Omeprazole 40 mg and dexamethasone 4 mg will be administered before the procedure as standard internal practice.

In the THRIVE group, dedicated Optiflow THRIVETM nasal cannulas will be positioned for 100% high flow oxygen therapy at an initial flow of 30 L/min. After induction of anesthesia and throughout the procedure the flow of oxygen will be increased to 70 L/min.

In the control group (CONTROL) after induction of anesthesia the patient will be mechanically ventilated through an I-Gel laryngeal mask.

General anesthesia, as per normal clinical practice, will be induced and maintained by target-controlled infusion (TCI) of propofol (7 mcg/Kg) by Orchestra Infusion system (Fresenius Kabi) and fentanyl 1.5 mcg/kg and in both groups. Propofol infusion rate will be between 3-4 mcg/ml for propofol, so to maintain a level of sedation monitored via BIS between 40-50. Paracetamol 1g, ondansetron 4 mg and ketorolac 30 mg will also be administered as per normal clinical practice.

In case of desaturation episodes, defined as a SpO2< 94% or increases in tcCO2 above 65 mmHg, the patient will be assisted with positive pressure ventilation through a facial or laryngeal mask or oro-tracheal intubation based on clinical judgment of the anesthesiologist.

At the end of the hysteroscopy the patient will be transferred to the Post-Anesthesia Care Unit (PACU) for 3 hours of post-procedural monitoring as required by internal protocol for day-surgery procedures. Standard monitoring will include non-invasive, intermittent (every 15 minutes) blood pressure monitoring, 3-leads electrocardiogram and peripheral oxygen saturation (SpO2).

One hour after the end of the procedure and before discharge from the PACU the patient will be asked to quantify the perceived degree of dyspnea with the Borg dyspnoea score and the degree of comfort using a Visual Numeric Scale (VAS) ranging from 0 to 10. In case of SpO2<94%, additional oxygen will be administered by means of a Venturi-type face mask with FiO2 40%. Discharge from the PACU will require an Aldrete score of 9-10.

Statistics The data will be analyzed according to an intention-to-treat principle. Clinical and demographic characteristics of the sample will be described through descriptive statistical techniques. Continuous quantitative variables with normal distribution will be reported as mean and standard deviation; as median and interquartile range the non-normal variables.

Categorical variables and missing data will be presented as absolute values and percentage, n (%).

Continuous variables will be compared with the Student t-test in case of normal distribution or, if not, with the Mann-Whitney test for independent samples. The normality of the distribution of the variables will be verified graphically by histograms and with the Shapiro-Wilk test.

Continuous variables with repeated measurements will be compared with a mixed-effect linear regression model. The type of airway management used and the timing at which the measurements will be performed will be considered as fixed effects; a random effect related to the patient will also be added.

The assumption of normality of the residues of the model will be graphically verified by histograms and Q-Q plots. The P-values will be obtained with the likelihood ratio test of the complete model with the effect in question with respect to the model without the effect. The estimates of the predictors used in the model will be reported with the relative 95% confidence intervals and P-values obtained with the Wald test.

In case of failure of the technique, defined as a transcutaneous concentration of carbon dioxide (tcCO2) > 65 mmHg and/or SpO2 < 94% in any of the study groups, a time-to-event (Kaplan-Meier) analysis will be carried out that takes into account the different duration of the procedures and therefore the different risk ranges for the possible onset of hypercapnia and / hypoxemia.

Differences between categorical data will be reported in terms of relative risk or risk differences, 95% confidence intervals and p-values based on the Χ2 test or fisher's exact test.

The significance level will be set for α < 0.05. All analyses will be performed with the statistical software R version 4.1.2 (R Foundation for Statistical Computing, Austria).

Continuous variables with repeated measurements will be compared with a mixed-effect linear regression model. Normality of distribution will be verified with the Shapiro-Wilk test. Continuous variables will be compared with Student t - or Mann Whitney test; categorical variables with the Chi-square test.

Sample size calculation In 2021, Kim et al. compared the safety of high flow oxygen therapy to conventional low-flow oxygen support for gastrointestinal endoscopic procedures performed under sedation reporting minimum values of peripheral saturation detected by pulse-oximeter higher in the high-flow group (99.8%) compared to low-flow oxygen therapy (95.1%).

To our knowledge, no study has compared these two methods during operative hysteroscopies under procedural sedation.

Based on literature and on the results from an internal registered pilot study in which we investigated the success rate of THRIVE as unique airway management technique in this setting, assuming a similar success rate of 95% for THRIVE and laryngeal mask ventilation, for a unilateral confidence interval of 95% and a 90% test power, we estimated a minimum sample of 82 patients per group to test a non-inferiority limit of 10%. The sample was increased to 90 patients for group to take into account any dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing operative hysteroscopy
* ASA I-II.

Exclusion Criteria:

* BMI > 30,
* pregnancy,
* cardiac arrhythmia,
* high risk of aspiration,
* neuromuscular disease,
* patient refusal.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of success of ventilation with THRIVE. | Throughout the surgical procedure
  Comparison of the rate of success in airways management with the THRIVE system versus positive pressure ventilation by laryngeal mask.
  The failure of the method will be defined as a CO2 value measured by transcutaneous monitor (Radiometer) > 65 mmHg AND/OR a peripheral O2 saturation measured by pulse oximeter < 94%.

SECONDARY OUTCOMES:
Airway related complications. | At the end of the surgery.
  Comparison of percentage of patients requiring airway manipulations (nasal cannula, manual ventilation, laryngeal mask ventilation, tracheal intubation) by the anesthesiologist in the two groups
Postoperative complications - 1 | At the end of the surgery.
  Comparison of percentage of patients suffering from cough, sore throat, dysphagia, dysphonia, laryngospasm, oxygen desaturation (defined as SpO2<94%).
Postoperative complications - 2 | At the end of the surgery.
  Comparison of incidence of dyspnoea (measured with Borg dyspnoea score: 0= no dyspnoea, 10= maximal dyspnoea) in the two groups.
Postoperative complications - 3 | At the end of the surgery.
  Comparison of incidence of discomfort (measured with Visual Analogue Scale: 0= no discomfort, 10= maximal discomfort) in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Policlinico A. Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] BARTLETT RG Jr, BRUBACH HF, SPECHT H. Demonstration of aventilatory mass flow during ventilation and apnea in man. J Appl Physiol. 1959 Jan;14(1):97-101. doi: 10.1152/jappl.1959.14.1.97. No abstract available. PMID 13630833
- [Result] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Result] O'Cain CF, Dowling NB, Slutsky AS, Hensley MJ, Strohl KP, McFadden ER Jr, Ingram RH Jr. Airway effects of respiratory heat loss in normal subjects. J Appl Physiol Respir Environ Exerc Physiol. 1980 Nov;49(5):875-80. doi: 10.1152/jappl.1980.49.5.875. PMID 7429910
- [Result] Slutsky AS, Brown R. Cardiogenic oscillations: a potential mechanism enhancing oxygenation during apneic respiration. Med Hypotheses. 1982 Apr;8(4):393-400. doi: 10.1016/0306-9877(82)90032-9. PMID 6808323
- [Result] Hermez LA, Spence CJ, Payton MJ, Nouraei SAR, Patel A, Barnes TH. A physiological study to determine the mechanism of carbon dioxide clearance during apnoea when using transnasal humidified rapid insufflation ventilatory exchange (THRIVE). Anaesthesia. 2019 Apr;74(4):441-449. doi: 10.1111/anae.14541. Epub 2019 Feb 15. PMID 30767199
- [Result] Brzek A, Dworrak T, Strauss M, Sanchis-Gomar F, Sabbah I, Dworrak B, Leischik R. The weight of pupils' schoolbags in early school age and its influence on body posture. BMC Musculoskelet Disord. 2017 Mar 21;18(1):117. doi: 10.1186/s12891-017-1462-z. PMID 28320364
- [Result] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Result] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405
- [Result] Parke RL, Bloch A, McGuinness SP. Effect of Very-High-Flow Nasal Therapy on Airway Pressure and End-Expiratory Lung Impedance in Healthy Volunteers. Respir Care. 2015 Oct;60(10):1397-403. doi: 10.4187/respcare.04028. Epub 2015 Sep 1. PMID 26329355
- [Result] Chikata Y, Onodera M, Oto J, Nishimura M. FIO2 in an Adult Model Simulating High-Flow Nasal Cannula Therapy. Respir Care. 2017 Feb;62(2):193-198. doi: 10.4187/respcare.04963. Epub 2016 Nov 22. PMID 27879385
- [Result] Moller W, Feng S, Domanski U, Franke KJ, Celik G, Bartenstein P, Becker S, Meyer G, Schmid O, Eickelberg O, Tatkov S, Nilius G. Nasal high flow reduces dead space. J Appl Physiol (1985). 2017 Jan 1;122(1):191-197. doi: 10.1152/japplphysiol.00584.2016. Epub 2016 Nov 17. PMID 27856714
- [Result] Gustafsson IM, Lodenius A, Tunelli J, Ullman J, Jonsson Fagerlund M. Apnoeic oxygenation in adults under general anaesthesia using Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) - a physiological study. Br J Anaesth. 2017 Apr 1;118(4):610-617. doi: 10.1093/bja/aex036. PMID 28403407
- [Result] Wong DT, Dallaire A, Singh KP, Madhusudan P, Jackson T, Singh M, Wong J, Chung F. High-Flow Nasal Oxygen Improves Safe Apnea Time in Morbidly Obese Patients Undergoing General Anesthesia: A Randomized Controlled Trial. Anesth Analg. 2019 Oct;129(4):1130-1136. doi: 10.1213/ANE.0000000000003966. PMID 31584919
- [Result] Mazzeffi MA, Petrick KM, Magder L, Greenwald BD, Darwin P, Goldberg EM, Bigeleisen P, Chow JH, Anders M, Boyd CM, Kaplowitz JS, Sun K, Terrin M, Rock P. High-Flow Nasal Cannula Oxygen in Patients Having Anesthesia for Advanced Esophagogastroduodenoscopy: HIFLOW-ENDO, a Randomized Clinical Trial. Anesth Analg. 2021 Mar 1;132(3):743-751. doi: 10.1213/ANE.0000000000004837. PMID 32398433
- [Result] Shih CC, Liang PC, Chuang YH, Huang YJ, Lin PJ, Wu CY. Effects of high-flow nasal oxygen during prolonged deep sedation on postprocedural atelectasis: A randomised controlled trial. Eur J Anaesthesiol. 2020 Nov;37(11):1025-1031. doi: 10.1097/EJA.0000000000001324. PMID 32890016
- [Result] Itagaki T, Okuda N, Tsunano Y, Kohata H, Nakataki E, Onodera M, Imanaka H, Nishimura M. Effect of high-flow nasal cannula on thoraco-abdominal synchrony in adult critically ill patients. Respir Care. 2014 Jan;59(1):70-4. doi: 10.4187/respcare.02480. Epub 2013 Jun 4. PMID 23737548
- [Result] Kagan I, Hellerman-Itzhaki M, Neuman I, Glass YD, Singer P. Reflux events detected by multichannel bioimpedance smart feeding tube during high flow nasal cannula oxygen therapy and enteral feeding: First case report. J Crit Care. 2020 Dec;60:226-229. doi: 10.1016/j.jcrc.2020.08.005. Epub 2020 Aug 22. PMID 32882605
- [Result] Coudroy R, Frat JP, Ehrmann S, Pene F, Terzi N, Decavele M, Prat G, Garret C, Contou D, Bourenne J, Gacouin A, Girault C, Dellamonica J, Malacrino D, Labro G, Quenot JP, Herbland A, Jochmans S, Devaquet J, Benzekri D, Vivier E, Nseir S, Colin G, Thevenin D, Grasselli G, Assefi M, Guerin C, Bougon D, Lherm T, Kouatchet A, Ragot S, Thille AW; REVA Network. High-flow nasal oxygen therapy alone or with non-invasive ventilation in immunocompromised patients admitted to ICU for acute hypoxemic respiratory failure: the randomised multicentre controlled FLORALI-IM protocol. BMJ Open. 2019 Aug 10;9(8):e029798. doi: 10.1136/bmjopen-2019-029798. PMID 31401603
- [Result] Mauri T, Galazzi A, Binda F, Masciopinto L, Corcione N, Carlesso E, Lazzeri M, Spinelli E, Tubiolo D, Volta CA, Adamini I, Pesenti A, Grasselli G. Impact of flow and temperature on patient comfort during respiratory support by high-flow nasal cannula. Crit Care. 2018 May 9;22(1):120. doi: 10.1186/s13054-018-2039-4. PMID 29743098
- [Derived] Frassanito L, Grieco DL, Vassalli F, Piersanti A, Scorzoni M, Ciano F, Zanfini BA, Catarci S, Catena U, Scambia G, Antonelli M, Draisci G. High-Flow Nasal Oxygen versus Mechanical Ventilation Through a Laryngeal Mask During General Anesthesia Without Muscle Paralysis: A Randomized Clinical Trial. Anesth Analg. 2025 Nov 1;141(5):1116-1125. doi: 10.1213/ANE.0000000000007620. Epub 2025 Jul 21. PMID 40690380